CLINICAL TRIAL: NCT02114359
Title: Comparison of Efficacy and Tolerance Between Combination Therapy and Monotherapy as a First Line Chemotherapy in Elderly Patient With Advanced Gastric Cancer; Multicenter Randomized Phase 3 Study
Brief Title: Chemotherapy Options for the First Line Chemotherapy in Elderly Patient With Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, In Sil Choi, Clinical Associate Professor, Department of Internal Medicine, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140113/16-2014-9/021
Record Dates: First submitted 2014-04-09; First posted 2014-04-15 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, elderly, chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Cisplatin; S-1 plus cisplatin; XELOX; Fluorouracil; Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platinum/fluoropyrimidine combination chemotherapy (Experimental)
  Interventions: Drug: Capecitabine/cisplatin; Drug: S-1/cisplatin; Drug: Capecitabine/oxaliplatin; Drug: 5-fluorouracil/oxaliplatin
- Fluoropyrimidine monochemotherapy (Active Comparator)
  Interventions: Drug: Capecitabine; Drug: S-1; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Capecitabine/cisplatin — Capecitabine/cisplatin (XP) : cisplatin 50mg/m2 (80% dose of 60mg/2m) iv over 15min D1, capecitabine 1000mg/m2 (80% dose of 1250mg/m2) po bid D1-14, q 3wks
  Arms: Platinum/fluoropyrimidine combination chemotherapy
Drug: S-1/cisplatin — S-1/cisplatin (SP) : cisplatin 50mg/m2 (80% dose of 60mg/2m) iv ov 15min D1, S-1 30mg/m2 (80% dose of 40mg/m2) po bid D1-14, q3wks
  Arms: Platinum/fluoropyrimidine combination chemotherapy
Drug: Capecitabine/oxaliplatin — Capecitabine+oxaliplatin (XELOX): oxaliplatin 100mg/m2 (80% dose of 130mg/m2)iv ov 120min D1, capecitabine 800mg/m2 (80% dose of 1000mg/m2) po bid D1-14, q3wks
  Arms: Platinum/fluoropyrimidine combination chemotherapy
Drug: 5-fluorouracil/oxaliplatin — 5-fluorouracil/oxaliplatin (FOLFOX): oxaliplatin 80mg/m2 (80% dose of 100mg/m2) iv ov 120min, leucovorin 80mg/m2 (80% dose of 100mg/m2) iv ov 120min, 5-fluorouracil 1900mg/m2 (80% dose of 2400mg/m2) iv ov 46h D1, q 2wks
  Arms: Platinum/fluoropyrimidine combination chemotherapy
Drug: Capecitabine — Capecitabine : 1250mg/m2 po bid D1-14 q3wks (if Ccr <60ml/min, 1000mg/m2 po bid)
  Arms: Fluoropyrimidine monochemotherapy
Drug: S-1 — S-1 : 40mg/m2 po bid D1-14 q3wks (if Ccr <60ml/min, 30mg/m2 po bid)
  Arms: Fluoropyrimidine monochemotherapy
Drug: 5-fluorouracil — 5-fluorouracil (FL) : leucovorin 100mg/m2 iv ov 2h, 5-fluorouracil 2400mg/m2 iv ov 46h D1, q2wks
  Arms: Fluoropyrimidine monochemotherapy

SUMMARY:
The investigators compare the overall survival between combination chemotherapy and monochemotherapy as a first-line chemotherapy in elderly patients with metastatic or recurrent gastric cancer. The investigators also compare the progression free survival, response rate, safety, and, quality of life between two groups, and evaluate that the comprehensive geriatric assessment tested at baseline can predict the toxicity and compliance of treatment, survival of the patients.

ELIGIBILITY:
Inclusion Criteria:

* .Metastatic or recurrent, histologically confirmed adenocarcinoma of stomach - Previously untreated patients, including patients with previous adjuvant chemotherapy completed more than 6 months
* 70 yrs or older
* Eastern Cooperative Oncology Group 0-2
* Measurable or evaluable disease
* Adequate major organ functions

  * Hb ≥ 9.0 g/dL
  * White blood cell count ≥ 3000/μL
  * Absolute Neutrophil Count (ANC) ≥ 1500/μL [*ANC = neutrophil segs ＋ neutrophil bands]
  * Platelet ≥ 100 × 103/ μL
  * Total bilirubin ≤ 1.5 ×UNL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3.0x UNL(in case of liver metastasis, AST/ALT ≤ 5.0 x UNL)
  * Serum creatinine ≤ 1.5 × UNL (in case of serum creatinine > 1.5 mg/dL , Ccr should be >= 50 mL/min, Ccr is calculated by Cockcroft-Gault or 24hr urine collection)
* Life expectancy > 3month
* Written informed consent

Exclusion Criteria:

* Metastatic or recurrent stomach cancer other than adenocarcinoma
* HER-2 positive
* Clinically significant, uncontrolled gastric outlet obstruction, bleeding, or perforation
* Radiation therapy within the previous 2wks
* Major surgery or trauma within the previous 4wks
* Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix)
* Uncontrolled brain metastasis
* Presence of other serious disease (cardiovascular, hepatic, infection etc.)
* Patients who participated in other clinical trials within the previous 30days
* Men of childbearing potential not willing to use effective means of contraception

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-02; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
comparison of overall survival | upto 3years

SECONDARY OUTCOMES:
comparison of progression-free survival | upto 2years
comparison of response rate | upto 2years
comparison of adverse events | upto 2yrs
comparison of quality of life | upto 2years

OTHER OUTCOMES:
comprehensive geriatric assessment | baseline
  The investigators are going to evaluate that comprehensive geriatric assessment tested at baseline can predict the toxicity and compliance to treatment, survival of patients.
  Comprehensive geriatric assessment will not necessarily be tested in all subjects, but instead, screening tool (KG-7 (Korean screening tool for the elderly)) will be tested in all subjects.

CONTACTS AND LOCATIONS:
Overall Officials: IN SIL CHOI, M.D., Ph.D., Principal Investigator — SMG-SNU Boramae Medical Center
Locations (14):
- South Korea (14):
  - Hallym University Sacred Heart Hospital, Anyang
  - Inje University Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Medical Center, Daegu
  - Yeongnam University Medical Center, Daegu
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Inje University Pusan Paik Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si

REFERENCES:
- [Background] Kim NK, Park YS, Heo DS, Suh C, Kim SY, Park KC, Kang YK, Shin DB, Kim HT, Kim HJ, et al. A phase III randomized study of 5-fluorouracil and cisplatin versus 5-fluorouracil, doxorubicin, and mitomycin C versus 5-fluorouracil alone in the treatment of advanced gastric cancer. Cancer. 1993 Jun 15;71(12):3813-8. doi: 10.1002/1097-0142(19930615)71:123.0.co;2-5. PMID 8508349
- [Background] Ohtsu A, Shimada Y, Shirao K, Boku N, Hyodo I, Saito H, Yamamichi N, Miyata Y, Ikeda N, Yamamoto S, Fukuda H, Yoshida S; Japan Clinical Oncology Group Study (JCOG9205). Randomized phase III trial of fluorouracil alone versus fluorouracil plus cisplatin versus uracil and tegafur plus mitomycin in patients with unresectable, advanced gastric cancer: The Japan Clinical Oncology Group Study (JCOG9205). J Clin Oncol. 2003 Jan 1;21(1):54-9. doi: 10.1200/JCO.2003.04.130. PMID 12506170
- [Background] Vanhoefer U, Rougier P, Wilke H, Ducreux MP, Lacave AJ, Van Cutsem E, Planker M, Santos JG, Piedbois P, Paillot B, Bodenstein H, Schmoll HJ, Bleiberg H, Nordlinger B, Couvreur ML, Baron B, Wils JA. Final results of a randomized phase III trial of sequential high-dose methotrexate, fluorouracil, and doxorubicin versus etoposide, leucovorin, and fluorouracil versus infusional fluorouracil and cisplatin in advanced gastric cancer: A trial of the European Organization for Research and Treatment of Cancer Gastrointestinal Tract Cancer Cooperative Group. J Clin Oncol. 2000 Jul;18(14):2648-57. doi: 10.1200/JCO.2000.18.14.2648. PMID 10894863
- [Background] Lacave AJ, Baron FJ, Anton LM, Estrada E, De Sande LM, Palacio I, Esteban E, Gracia JM, Buesa JM, Fernandez OA, et al. Combination chemotherapy with cisplatin and 5-fluorouracil 5-day infusion in the therapy of advanced gastric cancer: a phase II trial. Ann Oncol. 1991 Nov-Dec;2(10):751-4. doi: 10.1093/oxfordjournals.annonc.a057858. PMID 1801881
- [Background] Kang YK, Kang WK, Shin DB, Chen J, Xiong J, Wang J, Lichinitser M, Guan Z, Khasanov R, Zheng L, Philco-Salas M, Suarez T, Santamaria J, Forster G, McCloud PI. Capecitabine/cisplatin versus 5-fluorouracil/cisplatin as first-line therapy in patients with advanced gastric cancer: a randomised phase III noninferiority trial. Ann Oncol. 2009 Apr;20(4):666-73. doi: 10.1093/annonc/mdn717. Epub 2009 Jan 19. PMID 19153121
- [Background] Koizumi W, Narahara H, Hara T, Takagane A, Akiya T, Takagi M, Miyashita K, Nishizaki T, Kobayashi O, Takiyama W, Toh Y, Nagaie T, Takagi S, Yamamura Y, Yanaoka K, Orita H, Takeuchi M. S-1 plus cisplatin versus S-1 alone for first-line treatment of advanced gastric cancer (SPIRITS trial): a phase III trial. Lancet Oncol. 2008 Mar;9(3):215-21. doi: 10.1016/S1470-2045(08)70035-4. Epub 2008 Feb 20. PMID 18282805
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Lee JL, Kang YK, Kang HJ, Lee KH, Zang DY, Ryoo BY, Kim JG, Park SR, Kang WK, Shin DB, Ryu MH, Chang HM, Kim TW, Baek JH, Min YJ. A randomised multicentre phase II trial of capecitabine vs S-1 as first-line treatment in elderly patients with metastatic or recurrent unresectable gastric cancer. Br J Cancer. 2008 Aug 19;99(4):584-90. doi: 10.1038/sj.bjc.6604536. Epub 2008 Jul 29. PMID 18665164
- [Background] Koizumi W, Kurihara M, Nakano S, Hasegawa K. Phase II study of S-1, a novel oral derivative of 5-fluorouracil, in advanced gastric cancer. For the S-1 Cooperative Gastric Cancer Study Group. Oncology. 2000 Apr;58(3):191-7. doi: 10.1159/000012099. PMID 10765119